CLINICAL TRIAL: NCT01101958
Title: A Study of the Use of Chartis System to Optimize Subject Selection for Endobronchial Lung Volume Reduction (ELVR) in Subjects With Heterogeneous Emphysema
Brief Title: A Study of the Use of Chartis System to Optimize Subject Selection for Endobronchial Lung Volume Reduction (ELVR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulmonx Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 630-0011
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Results first posted 2014-01-23 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema | interventions — Therapeutics

ARMS (1):
- Chartis System-EBV Treatment (Other): Subjects with heterogeneous emphysema, had their collateral ventilation status in the target treatment lobe assessed using the Chartis System (CV- or CV+) and underwent endobronchial lung volume reduction (ELVR) with endobronchial valves (EBV).
  Interventions: Device: Chartis System; Device: Endobronchial Valve (EBV) Treatment

INTERVENTIONS:
Device: Chartis System — The Chartis System provides a value that represents the quantification of the average resistance to airflow through collateral airways.
Device: Endobronchial Valve (EBV) Treatment — The endobronchial valve is designed to induce target lobe volume reduction.

SUMMARY:
Use of the Chartis® Assessment System prior to EBV Treatment

DETAILED DESCRIPTION:
This is a multi-center study which will enroll up to 120 patients. Subjects will undergo a Chartis Assessment prior to EBV treatment. The Chartis assessment will determine the presence or absence of collateral ventilation, a potential determining factor in the success of EBV therapy. This study is not randomized; all subjects are eligible to receive EBV Treatment, regardless of Chartis Assessment outcome. Follow-up data will only be collected on those patients that meet the Chartis inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Heterogeneous emphysema
* Able to obtain a Chartis value during Assessment

Exclusion Criteria:

* Any co-existing major medical problems that would not make it possible for the subject to tolerate a bronchoscopic procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- University of Heidelberg, Heidelberg, Germany
- UMC Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Herth FJ, Eberhardt R, Gompelmann D, Ficker JH, Wagner M, Ek L, Schmidt B, Slebos DJ. Radiological and clinical outcomes of using Chartis to plan endobronchial valve treatment. Eur Respir J. 2013 Feb;41(2):302-8. doi: 10.1183/09031936.00015312. Epub 2012 May 3. PMID 22556025

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm--CV Negative: This arm was determined to have little or no collateral ventilation in the target treatment lobe as measured using the Chartis Pulmonary Assessment System.
- Treatment Arm--CV Positive: This arm was determined to have collateral ventilation in the target treatment lobe as measured using the Chartis Pulmonary Assessment System.
Period: Overall Study
Arm/Group | Treatment Arm--CV Negative | Treatment Arm--CV Positive
Started | 62 | 34
Completed | 51 | 29
Not Completed | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm--CV Negative: This arm had emphysema and was determined during bronchoscopy to have little or no collateral ventilation in the target treatment lobe as measured using the Chartis Pulmonary Assessment System.
- Treatment Arm--CV Positive: This arm had emphysema and was determined during bronchoscopy to have collateral ventilation in the target treatment lobe as measured using the Chartis Pulmonary Assessment System.
- Total: Total of all reporting groups
Arm/Group | Treatment Arm--CV Negative | Treatment Arm--CV Positive | Total
Number analyzed (Participants) | 62 | 34 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10) | 63 (9) | 63 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 19 | 49
  Male | 32 | 15 | 47
Region of Enrollment [Number; unit: participants]
  Netherlands | 21 | 9 | 30
  Germany | 34 | 23 | 57
  Sweden | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Lung Volume Change
Time Frame: 30 Days
Population: Per protocol population analyzed [16 subjects have been excluded due to the following reasons: lacked HRCT(n=6), Lost to Follow-Up (n=8) or died (n=2) of unrelated causes].
Measure: Median (Inter-Quartile Range); unit: percent decrease in lung volume
Arm/Group | Treatment Arm--CV Negative | Treatment Arm--CV Positive
Number analyzed (Participants) | 51 | 29
percent decrease in lung volume | 56 [18 to 92] | 6 [2 to 16]

ADVERSE EVENTS:
Arm/Group | Treatment Arm--CV Negative | Treatment Arm--CV Positive
Serious Adverse Events (participants affected / at risk) | 6/51 | 5/29
Other Adverse Events (participants affected / at risk) | 0/51 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm--CV Negative (N=51) | Treatment Arm--CV Positive (N=29)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less